CLINICAL TRIAL: NCT07151755
Title: Microneedle Intra-Arterial Injection With Pars Plana Vitrectomy for Acute Retinal Artery Occlusion: A Prospective Clinical Trial
Brief Title: Microneedle Intra-Arterial Injection for Retinal Artery Occlusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20251159
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Central Retinal Artery Occlusion
Keywords: central retinal artery occlusion; microneedle; thrombolysis
MeSH Terms: conditions — Retinal Artery Occlusion | interventions — Vitrectomy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitrectomy + Direct Intra-Arterial Microneedle Thrombolysis + Standard Care (Experimental): The patients will receive standard pars plana vitrectomy (PPV) combined with direct intra-arterial microneedle thrombolysis under microscopic visualization, in addition to standard clinical treatment for RAO. A 47G microneedle will be used to deliver thrombolytic agent intra-arterially per protocol.
  Interventions: Procedure: Standard Clinical Care Only
- Standard Clinical Care Only (Active Comparator): The patients will receive standard clinical treatment for RAO without vitrectomy or intra-arterial microneedle thrombolysis.
  Interventions: Procedure: Vitrectomy + Direct Intra-Arterial Microneedle Thrombolysis + Standard Care

INTERVENTIONS:
Procedure: Vitrectomy + Direct Intra-Arterial Microneedle Thrombolysis + Standard Care — The patients will receive standard pars plana vitrectomy (PPV) combined with direct intra-arterial microneedle thrombolysis under microscopic visualization, in addition to standard clinical treatment for RAO. A 47G microneedle will be used to deliver thrombolytic agent intra-arterially per protocol.
  Arms: Standard Clinical Care Only
Procedure: Standard Clinical Care Only — The patients will receive standard clinical treatment for RAO without vitrectomy or intra-arterial microneedle thrombolysis.
  Arms: Vitrectomy + Direct Intra-Arterial Microneedle Thrombolysis + Standard Care

SUMMARY:
This prospective interventional study evaluates the efficacy and safety of direct intra-arterial microneedle injection combined with pars plana vitrectomy for acute retinal artery occlusion (including central retinal artery occlusion [CRAO] and branch retinal artery occlusion [BRAO] involving the macula or causing severe visual loss). The primary endpoint is best-corrected visual acuity (BCVA, LogMAR) at 1 month. Secondary objectives include assessing the effect of treatment timing and monitoring longitudinal changes in visual function and retinal structure over 12 months.

DETAILED DESCRIPTION:
Retinal artery occlusion lacks an established standard therapy. This prospective, non-randomized, parallel-group interventional trial compares pars plana vitrectomy with direct intra-arterial microneedle thrombolysis plus standard care (experimental arm) with standard clinical care alone (control arm). The trial is open-label, and outcome assessors for BCVA, automated perimetry, fluorescein angiography (FFA), and optical coherence tomography (OCT) will be masked. Scheduled visits occur at 1 week, 1 month, 3 months, 6 months, and 12 months. The symptom-to-treatment interval (≤3 days vs 3-7 days) is a prespecified subgroup for secondary analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute non-arteritic retinal artery occlusion (RAO), including: Central retinal artery occlusion (CRAO), or Branch retinal artery occlusion (BRAO) involving the macula or causing severe visual loss; defined as symptom onset ≤7 days and confirmed by exam ± imaging (FFA/OCT)
* Best-corrected visual acuity (BCVA) <0.5 (decimal)

Exclusion Criteria:

* Active bleeding disorder, or significant bleeding within the past 3 months, or bleeding diathesis
* Severe hypertension: SBP >185 mmHg or DBP >110 mmHg
* Severe coagulopathy or ongoing therapeutic anticoagulation
* Ischemic stroke within the past 3 months
* Severe, unstable systemic disease rendering surgery or anesthesia risk unacceptable
* Known hypersensitivity to thrombolytic agents or any study medications/materials
* Active ocular infection
* Vitreous hemorrhage
* Retinal arteritis
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Best-Corrected Visual Acuity | 1 month postoperatively

SECONDARY OUTCOMES:
Visual Field Improvement | Baseline to 1 week, 1, 3, 6, and 12 months postoperatively
  Humphrey Perimetry
Retinal Reperfusion Rate | Baseline to 1 week, 1, 3, 6, and 12 months postoperatively
  fluorescein fundus angiography
OCT/OCTA Structural-Perfusion Changes | Baseline to 1 week, 1, 3, 6, and 12 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Center of the Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No